CLINICAL TRIAL: NCT05164237
Title: Multimodal Approach of Electrotherapy Versus Nerve Flossing Technique in Patient With Carpal Tunnel Syndrome
Acronym: CTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, heba Haridy, assistant lecturer, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 85632
Record Dates: First submitted 2021-12-05; First posted 2021-12-20 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Experimental): 17 subjects will receive multimodal approach of electrotherapy (LLLT , US and IFC) with conventional physical therapy modalities in the form of ( splint and therapeutic exercises ) 3 sessions every week for 8 weeks.
  Interventions: Other: multimodal electrotherapy
- group B (Experimental): 17 subjects will receive NFT with conventional physical therapy modalities in the form of (splint and therapeutic exercises ) 3 sessions every week for 8 weeks.
  Interventions: Other: nerve flossing technique
- group C (Experimental): 17 subjects will receive with conventional physical therapy modalities only in the form of (splint and therapeutic exercises ) 3 sessions every week for 8 weeks.
  Interventions: Other: exercises

INTERVENTIONS:
Other: nerve flossing technique — subjects will receive NFT with conventional physical therapy modalities in the form of (splint and therapeutic exercises ) 3 sessions every week for 8 weeks.
  Arms: group B
Other: multimodal electrotherapy — subjects will receive multimodal approach of electrotherapy (LLLT , US and IFC) with conventional physical therapy modalities in the form of ( splint and therapeutic exercises ) 3 sessions every week for 8 weeks.
  Arms: group A
Other: exercises — subjects will receive with conventional physical therapy modalities only in the form of (splint and therapeutic exercises ) 3 sessions every week for 8 weeks.
  Arms: group C

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common and median nerve neuropathy at the wrist, caused by compression of the median nerve at the level of the carpal tunnel (CT) delimitated by the carpal bones and the transverse carpal ligament(TCL) which is the intermediate part of the flexor retinaculum (FR).

The CTS remains a challenge for health care providers due to its high prevalence and economic consequences, it is projected that in every 5 patients, 1 complains of symptoms of pain, numbness and a tingling sensation in the hands, CTS is estimated to occur in 3.8% of the general population with an incidence rate of 276:100000 per year and happens more frequently in women than in men so a prevalence rate of 9.2% in women and 6% in men

DETAILED DESCRIPTION:
The CTS is a common clinical problem caused by the entrapment of the median nerve at the wrist, It is an important mononeuropathy that causes of hand pain, neurologic symptoms, and functional limitation of the hand, It is the most common nerve compression disorder of the upper extremity ,it accounting for 90% of all neuropathies, It is estimated that CTS affects approximately is between 3.7% and 5.8% of the general population with a prevalence rate up to 9.2% in women and 6% in men , CTS is 10 times more frequent in women than men , the peak age range of CTS is between 40 to 60 years ,it is mostly seen in women ages between 30 to 50 years due to the housework they do, however, it occurs in all age groups

ELIGIBILITY:
Inclusion Criteria:

Fifty one female patients have unilateral with mild to moderate CTS in dominant hand diagnosed and reffered by physician.

Age will be ranged from 30-45years (Atya et al.,2020) Patients with mild to moderate CTS will particiepate into the current study according to the classification of AAEM

Exclusion Criteria:

Patients with diabetes mellities ( type I or type II), Patients with Hypertension Patients with hypothyroidism Patients with rheumatological disease Patients with renal disease

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Weight and height scale | 8 weeks
  Weighting scale will administreted by using (SH-8024) , it will be used to measure weight in kg and height in cm , of all patients before starting the assessment for determining BMI
Visual analogue scale | 8 weeks
  The VAS consists of a 10-cm line, with the left extremity indicating ''no pain'' and the right extremity indicating ''unbearable pain.'' Participants asked to use the scale to indicate their current level of pain Higher values suggest more intense pain ,It was found that VAS provide valid and reliable assessments for the affective magnitude, as well as the sensation intensity of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Heba, Cairo, Egypt